CLINICAL TRIAL: NCT01767038
Title: Study of Anatomical and Functional Recovery Following Retinal Detachment: Identify Correlations Between Visual Acuity and SD-OCT and Microperimetry Findings.
Brief Title: DOREFA (Retinal Detachment: Function and Anatomy)
Acronym: DOREFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Creuzot-Garcher PHRC N 2010
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: OCT Spectralis
Procedure: microperimetry

SUMMARY:
Patients with retinal detachment do not always recover good visual function. Sometimes simple causes are responsible. Other causes can only be discovered thanks to high-resolution imaging provided by the latest generation of OCT.

This study is possible thanks to surgical teams who have a strong recruitment potential, with the experience of a joint project in 2007-2008 (PHRC national - Etude DOREMY, Etude FRIENDS) to define more strict intervention criteria. The principal objective of this study is to better define with regard to time:

* The onset of surgically curable or transient macular affections, and losses in visual acuity that can be qualified as "explained"
* But above all to better understand the relationships between anatomical analyses obtained using OCT and autofluorescence and functional analysis using visual acuity and microperimetry.
* In the near future, two techniques (OCT and microperimetry) will certainly become essential tools in the evaluation of macular function. Better understanding of these relationships is the first necessary step in any study concerning the therapeutic prevention of retinal lesions related to retinal detachment: This study will make it possible to define criteria for the evaluation of anatomical and functional recovery, their relationship with each other and finally their evolution over time. This is an essential first phase before possible therapies can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written informed consent
* Retinal detachment with pre-operative raised macula, re-attached during a surgical intervention with one month of follow-up
* Patients undergoing surgery as the first-line treatment (ab extern surgery or gas vitrectomy)
* Patients who accept to be followed for at least 12 months at the investigating center.

Exclusion Criteria:

* Persons who are not registered with social security agency
* Macular affections pre-existent to the DR
* Retinal detachment requiring several interventions to obtain a reapplication
* Lazy eye with pre-operative
* Brightness of the circles not allowing the realization of the examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Relationship between functional recovery and the aspect of external layers using Spectral Domain OCT. | At six months after the intervention
  Visual acuity, integrity of the IS/OS junction of the photoreceptors and the outer limiting membrane.

SECONDARY OUTCOMES:
Peripheral deficits and quantification of hypoautofluorescent zones. | At 3, 6 and 12 months after intervention

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hôpital Lariboisière, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - CHU Reims - Hôpital Robert Debré, Reims
  - CHU Strasbourg - Hôpital Civil, Strasbourg

REFERENCES:
- [Result] Baudin F, Deschasse C, Gabrielle PH, Berrod JP, Le Mer Y, Arndt C, Tadayoni R, Delyfer MN, Weber M, Gaucher D, Saleh M, Chiquet C, Creuzot-Garcher C. Functional and anatomical outcomes after successful repair of macula-off retinal detachment: a 12-month follow-up of the DOREFA study. Acta Ophthalmol. 2021 Nov;99(7):e1190-e1197. doi: 10.1111/aos.14777. Epub 2021 Feb 11. PMID 33576133